CLINICAL TRIAL: NCT03400800
Title: A Placebo-Controlled, Double-Blind, Randomized Trial to Evaluate the Effect of 300 mg of Inclisiran Sodium Given as Subcutaneous Injections in Subjects With Atherosclerotic Cardiovascular Disease (ASCVD) or ACSVD Risk-Equivalents and Elevated Low-Density Lipoprotein Cholesterol (LDL-C)
Brief Title: Inclisiran for Subjects With ASCVD or ASCVD-Risk Equivalents and Elevated Low-density Lipoprotein Cholesterol
Acronym: ORION-11
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDCO-PCS-17-08
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Results first posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: ASCVD; Risk Factor, Cardiovascular; Elevated Cholesterol
Keywords: Inclisiran sodium; ASCVD; LDL-C
MeSH Terms: conditions — Hypercholesterolemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran (Experimental): Inclisiran sodium 300 milligrams (mg) (equivalent to 284 mg inclisiran) in 1.5 milliliters (mL) will be administered as a SC injection on Day 1, Day 90, and then every 6 months.
  Interventions: Drug: Inclisiran Sodium
- Saline Solution (Placebo Comparator): Placebo (1.5 mL) will be administered as a SC injection of saline solution on Day 1, Day 90, and then every 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclisiran Sodium — Inclisiran is a small interfering ribonucleic acid (RNA) that inhibits PCSK9 synthesis.
  Arms: Inclisiran
Drug: Placebo — Placebo will be supplied as sterile normal saline (0.9% sodium chloride in water for injection).
  Other Names: Saline Solution
  Arms: Saline Solution

SUMMARY:
This is a Phase III, placebo-controlled, double-blind, randomized study in participants with ASCVD or ASCVD-Risk equivalents and elevated LDL-C despite maximum tolerated dose of LDL-C lowering therapies to evaluate the efficacy, safety, and tolerability of subcutaneous (SC) inclisiran injection(s). The study will be an international multicenter study (non-United States).

ELIGIBILITY:
Inclusion Criteria:

Participants may be included if they meet all of the following inclusion criteria prior to randomization:

1. Male or female participants ≥18 years of age.
2. History of ASCVD (coronary heart disease [CHD], cardiovascular disease [CVD], or peripheral arterial disease [PAD]).
3. Serum LDL-C ≥1.8 millimole (mmol)/liter (L) (≥70 mg/dL).
4. Fasting triglyceride <4.52 mmol/L (<400 mg/dL) at screening.
5. Calculated glomerular filtration rate >30 mL/min by estimated glomerular filtration rate (eGFR) using standardized clinical methodology
6. Participants on statins should be receiving a maximally tolerated dose.
7. Participants not receiving statins must have documented evidence of intolerance to all doses of at least 2 different statins.
8. Subjects on lipid-lower therapies (such as a statin and/or ezetimibe) should be on a stable dose for ≥30 days before screening with no planned medication or dose change during study participation.
9. Subjects were willing and able to give informed consent before initiation of any study-related procedures and willing to comply with all required study procedures

Exclusion Criteria:

Participants will be excluded from the study if any of the following exclusion criteria apply prior to randomization:

1. New York Heart Association (NYHA) class IV heart failure.
2. Uncontrolled cardiac arrhythmia.
3. Uncontrolled severe hypertension.
4. Active liver disease.
5. Females who are pregnant or nursing, or who are of childbearing potential and unwilling to use at least 2 methods of highly effective contraception (failure rate less than 1% per year) (for example, combined oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, or intrauterine device) for the entire duration of the study. Exemptions from this criterion:

   1. Women >2 years postmenopausal (defined as 1 year or longer since last menstrual period) and more than 55 years of age.
   2. Postmenopausal women (as defined above) and less than 55 years of age with a negative pregnancy test within 24 hours of randomization.
   3. Women who are surgically sterilized at least 3 months prior to enrollment.
6. Males who are unwilling to use an acceptable method of birth control during the entire study period (such as condom with spermicide).
7. Treatment with other investigational products or devices within 30 days or 5 half-lives of the screening visit, whichever is longer.
8. Treatment (within 90 days of screening) with monoclonal antibodies directed towards PCSK9.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1617 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray Kausik, MD, Principal Investigator — Imperial College of London
Locations (70):
- Czechia (2):
  - Research Site 11420-002, Chomutov
  - Research Site 11420-003, Uherské Hradiště
- Germany (5):
  - Research Site 11049-006, Berlin
  - Research Site 11049-002, Bochum
  - Research Site 11049-003, Frankfurt
  - Research Site 11049-007, Heidelberg
  - Research Site 11049-001, Leipzig
- Hungary (4):
  - Research Site 11036-001, Budapest
  - Research Site 11036-004, Debrecen
  - Research Site 11036-002, Hatvan
  - Research Site 11036-003, Zalaegerszeg
- Poland (19):
  - Research Site 11048-018, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Research Site 11048-016, Brzozów, Podkarpackie Voivodeship
  - Research Site 11048-019, Ruda Śląska, Silesian Voivodeship
  - Research Site 11048-011, Bydgoszcz
  - Research Site 11048-004, Gdansk
  - Research Site 11048-017, Gdansk
  - Research Site 11048-005, Gdynia
  - Research Site 11048-007, Katowice
  - Research Site 11048-012, Katowice
  - Research Site 11048-014, Krakow
  - Research Site 11048-003, Krakow
  - Research Site 11048-008, Lublin
  - Research Site 11048-001, Poznan
  - Research Site 11048-013, Rzeszów
  - Research Site 11048-015, Tarnów
  - Research Site 11048-009, Warsaw
  - Research Site 11048-006, Warszawice
  - Research Site 11048-002, Wroclaw
  - Research Site 11048-010, Wroclaw
- South Africa (8):
  - Research Site 11027-003, Bloemfontein, Free State
  - Research Site 11027-005, Johannesburg, Gauteng
  - Research Site 11027-001, Cape Town, Western Cape
  - Research Site 11027-013, Cape Town, Western Cape
  - Research Site 11027-007, Kuils River, Western Cape
  - Research Site 11027-004, Somerset West, Western Cape
  - Research Site 11027-006, Pretoria
  - Research Site 11027-011, Welkom
- Ukraine (9):
  - Research Site - 11380-005, Cherkasy
  - Research Site - 11380-008, Kharkiv
  - Research Site - 11380-004, Kiev
  - Research Site - 11380-009, Kiev
  - Research Site - 11380-001, Kyiv
  - Research Site - 11380-002, Kyiv
  - Research Site - 11380-003, Kyiv
  - Research Site - 11380-007, Lviv
  - Research Site - 11380-006, Uzhhorod
- United Kingdom (23):
  - Research Site - 11044-006, Edgbaston, Birmingham
  - Research Site - 11044-022, Sale, Cheshire
  - Research Site - 11044-023, Sale, Cheshire
  - Research Site - 11044-021, Timperley, Cheshire
  - Research Site - 11044-012, Liskeard, Cornwall
  - Research Site - 11044-009, Exeter, Devon
  - Research Site - 11044-019, Plymouth, Devon
  - Research Site - 11044-014, Chorley, Lancashire
  - Research Site - 11044-004, Waterloo, Liverpool
  - Research Site - 11044-027, Davyhulme, Manchester
  - Research Site - 11044-028, Bollington
  - Research Site - 11044-026, Bury
  - Research Site - 11044-007, Cardiff
  - Research Site - 11044-024, Cheadle Hulme
  - Research Site - 11044-010, Derby
  - Research Site - 11044-001, Glasgow
  - Research Site - 11044-008, Hexham
  - Research Site - 11044-020, Macclesfield
  - Research Site - 11044-025, Manchester
  - Research Site - 11044-005, Manchester
  - Research Site - 11044-029, Manchester
  - Research Site - 11044-003, Reading
  - Research Site - 11044-002, Stockton

REFERENCES:
- [Derived] Wright RS, Ray KK, Landmesser U, Koenig W, Raal FJ, Leiter LA, Conde LG, Han J, Schwartz GG. Effects of Inclisiran in Patients With Atherosclerotic Cardiovascular Disease: A Pooled Analysis of the ORION-10 and ORION-11 Randomized Trials. Mayo Clin Proc. 2024 Jul 5:S0025-6196(24)00167-8. doi: 10.1016/j.mayocp.2024.03.025. Online ahead of print. PMID 39093262
- [Derived] Dutta S, Shah R, Singhal S, Singh S, Piparva K, Katoch CDS. A systematic review and meta-analysis of tolerability, cardiac safety and efficacy of inclisiran for the therapy of hyperlipidemic patients. Expert Opin Drug Saf. 2024 Feb;23(2):187-198. doi: 10.1080/14740338.2023.2293201. Epub 2023 Dec 19. PMID 38063346
- [Derived] Ray KK, Wright RS. Plain language summary of results from ORION-10 and ORION-11: two studies to learn how well inclisiran works in people with high cholesterol. Future Cardiol. 2023 Mar;19(4):175-184. doi: 10.2217/fca-2022-0133. Epub 2023 Jun 6. PMID 37282500
- [Derived] Ray KK, Wright RS, Kallend D, Koenig W, Leiter LA, Raal FJ, Bisch JA, Richardson T, Jaros M, Wijngaard PLJ, Kastelein JJP; ORION-10 and ORION-11 Investigators. Two Phase 3 Trials of Inclisiran in Patients with Elevated LDL Cholesterol. N Engl J Med. 2020 Apr 16;382(16):1507-1519. doi: 10.1056/NEJMoa1912387. Epub 2020 Mar 18. PMID 32187462

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (1.5 mL) will be administered as a SC injection of saline solution on Day 1, Day 90, and then every 6 months
  Placebo will be supplied as sterile normal saline (0.9% sodium chloride in water for injection).
Period: Overall Study
Arm/Group | Inclisiran | Placebo
Started | 810 | 807
Completed | 772 | 770
Not Completed | 38 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inclisiran | Placebo | Total
Number analyzed (Participants) | 810 | 807 | 1617
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 367 | 366 | 733
  >=65 years | 443 | 441 | 884
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (8.29) | 64.8 (8.68) | 64.8 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 231 | 226 | 457
  Male | 579 | 581 | 1160
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 12 | 8 | 20
  White | 791 | 796 | 1587
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 52 | 52 | 104
  Czechia | 10 | 11 | 21
  Ukraine | 55 | 54 | 109
  Poland | 360 | 357 | 717
  South Africa | 60 | 61 | 121
  United Kingdom | 231 | 231 | 462
  Germany | 42 | 41 | 83

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in LDL-C From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Inclisiran: Inclisiran sodium 300 milligrams (mg) (equivalent to 284 mg inclisiran) in 1.5 millilitres (mL) administered as a subcutaneous injection on Day 1, Day 90, and then every 6 months.
- Placebo: Placebo (1.5 mL) administered as a subcutaneous injection of sterile saline solution (0.9% sodium chloride in water for injection) on Day 1, Day 90, and then every 6 months.
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 810 | 807
Percent change | -49.3 [-51.22 to -47.48] | 4.2 [1.62 to 6.69]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -53.5, 95% CI 2-sided [-56.66 to -50.35] — Represents the least squares means difference from Placebo

2. Primary Outcome: Time-adjusted Percent Change in LDL-C Levels From Baseline After Day 90 and up to Day 540
Time Frame: Baseline, Day 90 to Day 540
Population: ITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 810 | 807
Percent change | -45.82 [-47.52 to -44.13] | 3.35 [1.65 to 5.05]
Statistical Analysis 1: Comparison: Inclisiran; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -49.17, 95% CI 2-sided [-51.57 to -46.77] — Represents the least squares means difference from Placebo

3. Secondary Outcome: Absolute Change In LDL-C From Baseline To Day 510
Time Frame: Baseline, Day 510
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 810 | 807
mg/dL | -50.91 [-53.14 to -48.67] | 0.96 [-1.26 to 3.18]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < .0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Median Difference (Final Values) = -51.87, 95% CI 2-sided [-55.01 to -48.72] — Represents the least squares means difference from Placebo

4. Secondary Outcome: Time-adjusted Absolute Change in LDL-C From Baseline After Day 90 and up to Day 540
Time Frame: Baseline, Day 90 to Day 540
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 810 | 807
mg/dL | -48.63 [-50.37 to -46.89] | 0.31 [-1.42 to 2.04]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -48.94, 95% CI 2-sided [-51.39 to -46.48] — Represents the least squares means difference from Placebo

5. Secondary Outcome: Percentage Change in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) From Baseline to Day 510
Time Frame: Baseline, Day 510
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 810 | 807
Percent change | -63.64 [-65.55 to -61.74] | 15.62 [13.72 to 17.53]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -79.27, 95% CI 2-sided [-81.97 to -76.57] — Represents the least squares means difference from Placebo

6. Secondary Outcome: Percentage Change in Total Cholesterol From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 810 | 807
Percent change | -28.00 [-29.40 to -26.60] | 1.79 [0.38 to 3.21]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -29.79, 95% CI 2-sided [-31.78 to -27.81] — Represents the least squares means difference from Placebo

7. Secondary Outcome: Percentage Change in Apolipoprotein B (ApoB) From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 810 | 807
Percent change | -38.15 [-39.76 to -36.54] | 0.79 [-0.82 to 2.41]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -38.94, 95% CI 2-sided [-41.21 to -36.67] — Represents the least squares means difference from Placebo

8. Secondary Outcome: Percentage Change in Non-HDL-C From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 810 | 807
Percent change | -41.16 [-43.09 to -39.24] | 2.15 [0.22 to 4.09]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -43.32, 95% CI 2-sided [-46.04 to -40.60] — Represents the least squares means difference from Placebo

ADVERSE EVENTS:
Time Frame: 17 months
Description: The Efficacy population was comprised of 807 (Placebo) and 810 (Inclisiran) for a toal of 1617 subjects. The Safety population consisted of 804 (Placebo) and 811 (Inclisiran). The reason for this discrepancy is because two randomized subjects (Placebo) were not dosed, so were randomized in error. In addition, a placebo subject received inclisiran at Day 450 so was reallocated into the inclisiran group for safety as per the definition.
Arm/Group | Inclisiran | Placebo
All-Cause Mortality (participants affected / at risk) | 14/811 | 15/804
Serious Adverse Events (participants affected / at risk) | 181/811 | 181/804
Other Adverse Events (participants affected / at risk) | 331/811 | 319/804
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=811) | Placebo (N=804)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 5 | 18
Angina pectoris (Cardiac disorders) | 14 | 13
Angina unstable (Cardiac disorders) | 11 | 11
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 10 | 6
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0
Cardiac failure (Cardiac disorders) | 3 | 6
Cardiac failure chronic (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 5 | 2
Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 8 | 11
Coronary artery insufficiency (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 5 | 4
Myocardial ischaemia (Cardiac disorders) | 4 | 5
Palpitations (Cardiac disorders) | 1 | 0
Paroxysmal arrhythmia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Silent myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hypopituitarism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 2
Large intestine polyp (Gastrointestinal disorders) | 1 | 2
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Cardiac death (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 2
Exercise tolerance decreased (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 4 | 8
Sudden cardiac death (General disorders) | 1 | 1
Vascular stent occlusion (General disorders) | 1 | 0
Vascular stent restenosis (General disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 3 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 2
Sarcoidosis (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 2 | 2
Biliary sepsis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 2 | 1
Chest wall abscess (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Gallbladder abscess (Infections and infestations) | 1 | 0
Gallbladder empyema (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 3
Neuroborreliosis (Infections and infestations) | 0 | 1
Pathogen resistance (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 9 | 7
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
Wound infection (Infections and infestations) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 0 | 1
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 0 | 1
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 3
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Undifferentiated connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Linitis plastica (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral nerve sheath tumour malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tracheal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain injury (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 3
Lacunar stroke (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 3 | 1
Device loosening (Product Issues) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
End stage renal disease (Renal and urinary disorders) | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 2
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0
Leg amputation (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 2
Aortic dissection (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Granulomatosis with polyangiitis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 0 | 1
Iliac artery embolism (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 7 | 8
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Thromboangiitis obliterans (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=811) | Placebo (N=804)
Nasopharyngitis (Infections and infestations) | 91 | 90
Upper respiratory tract infection (Infections and infestations) | 52 | 49
Diabetes mellitus (Metabolism and nutrition disorders) | 88 | 94
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 | 32
Hypertension (Vascular disorders) | 53 | 54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/00/NCT03400800/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT03400800/SAP_001.pdf